CLINICAL TRIAL: NCT01194453
Title: A Phase 2,Open-label Study of First Line Pemetrexed Plus Cisplatin Versus Gemcitabine Plus Cisplatin for Advanced and Metastatic Non Small Cell Lung Cancer and Biomarker Study
Brief Title: Pemetrexed Plus Cisplatin Versus Gemcitabine Plus Cisplatin for Advanced NSCLC Metastatic Non-small Cell Lung Cancer
Acronym: AP/GP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HANSOH20090601
Record Dates: First submitted 2010-08-25; First posted 2010-09-03 (Estimated); Results first posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: Non-small Cell Lung Cancer; Efficacy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Dexamethasone; Vitamin B 12; Folic Acid; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: cisplatin, dexamethasone,vitamin B12, folic acid
- Group B (Active Comparator)
  Interventions: Drug: cisplatin, gemcitabine

INTERVENTIONS:
Drug: cisplatin, dexamethasone,vitamin B12, folic acid — Patients received cisplatin 75mg/m2 plus pemetrexed 500 mg/m2 on day 1.Chemotherapy was repeated every 3 weeks for a maximum of six cycles.Patients received dexamethasone prophylaxis of 3.75mg orally twice per day on the day before, the day of, and the day after each day-1 treatment. patients received oral folic acid (1,000ug)daily and a vitamin B12 injection (1,000 ug) every 9 weeks, beginning 1 to 2 weeks before the first dose and continuing until 3 weeks after the last dose of study treatment
  Arms: Group A
Drug: cisplatin, gemcitabine — cisplatin 75mg/m2 on day 1 plus gemcitabine 1000 mg/m2 on days 1 and 8
  Arms: Group B

SUMMARY:
A phase III trial has demonstrated that in advanced non-small cell lung cancer (NSCLC) cisplatin/ pemetrexed provides similar efficacy with better tolerability and more convenient administration than cisplatin/gemcitabine. Moreover,this trial showed survival differences based on histologic type. The investigators want to research some biomarkers that can predict clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Chemotherapy-naive patients with histologically or cytologically confirmed adenocarcinoma and large-cell carcinoma, classified as stage IIIB not amenable to curative treatment or stage IV
2. With at least one unidimensionally measurable lesion according to the Response Evaluation Criteria in Solid Tumors;
3. with an Eastern CooperativeOncology Group performance status of 0 or 1,
4. At least 18 years of age
5. adequate bone marrow reserve and organ function including calculated creatinine clearance 45 mL/min based on the standard Cockcroft and Gault formula.
6. Prior radiation therapy was permitted if it was completed at least 4 weeks before study treatment
7. patients had fully recovered from its acute effects.

Exclusion Criteria:

1. peripheral neuropathy > National Cancer Institute Common Toxicity Criteria grade 1
2. progressive brain metastases,
3. uncontrolled third-space fluid retention before study entry.
4. Patients unable to interrupt aspirin and other nonsteroidal anti-inflammatory drugs or if they were unable or unwilling to take folic acid, vitamin B12, or corticosteroids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Study Chair — Cancer Center of Sun Yat-Sen University (CCSU)
Locations (1):
- Cancer Center of Sun Yat-Sen University (CCSU), Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Huang Y, Liu Y, Zhou J, Xu N, Li B, Wu G, Fang J, Li K, Liu X, Liu W, Lu Y, Wang M, Liu W, Liang H, Zhang Y, Huang C, Wang S, Wang Y, Yu S, Chang J, Wang Z, Hu Z, Zhang L. [A randomized, controlled, multicenter clinical trial comparing pemetrexed/cisplatin and gemcitabine/cisplatin as first-line treatment for advanced nonsquamous non-small cell lung cancer]. Zhongguo Fei Ai Za Zhi. 2012 Oct;15(10):576-82. doi: 10.3779/j.issn.1009-3419.2012.10.03. Chinese. PMID 23075681

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 144 | 144
Completed | 127 | 127
Not Completed | 17 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 144 | 144 | 288
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 129 | 120 | 249
  >=65 years | 15 | 24 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 73 | 133
  Male | 84 | 71 | 155
Region of Enrollment [Number; unit: participants]
  China | 144 | 144 | 288

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Time Frame: 36months
Measure: Median (95% Confidence Interval); unit: day
Arm/Group | Group A | Group B
Number analyzed (Participants) | 144 | 144
day | 168 [139 to 183] | 140 [113 to 164]

2. Secondary Outcome: Response Rate
Time Frame: 6 weeks
Measure: Number; unit: percentage
Arm/Group | Group A | Group B
Number analyzed (Participants) | 127 | 127
percentage | 24.41 | 14.17

ADVERSE EVENTS:
Time Frame: From the delivery of the study drug to 21 days post the last dose of study drug.
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 5/144 | 5/144
Other Adverse Events (participants affected / at risk) | 131/144 | 140/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=144) | Group B (N=144)
Leading to Hospitalization (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) — Obstructive pneumonia
Death (General disorders) | 1 (1) | 1 (1)
Life threatening (General disorders) | 1 (1) | 1 (1)
Delay hospitalization (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=144) | Group B (N=144)
leukopenia (Blood and lymphatic system disorders) | 63 (63) | 69 (69)
neutropenia (Blood and lymphatic system disorders) | 64 (64) | 59 (59)
anemia (Blood and lymphatic system disorders) | 34 (34) | 48 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No